CLINICAL TRIAL: NCT07207499
Title: Evaluation of the Access to Healthcare Service Established in the Le Havre Area
Brief Title: Evaluation of the Access to Healthcare Service
Acronym: SAS-LH
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0350/HP; 2023-A02103-42 (Other: ANSM)
Record Dates: First submitted 2025-09-26; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Emergency Service, Hospital
Keywords: Access to Care Service (SAS); telephone patient regulation service
MeSH Terms: conditions — Emergencies | interventions — Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: control group ("standard" regulation device) — Evaluate the time spent in the emergency room of patients referred to the emergency room by the "standard" regulation system
Other: intervention group Access to Care Service "SAS" — Evaluate the time spent in the emergency room of patients referred to the emergency room by the Emergency Care Access Service (SAS)

SUMMARY:
The Healthcare Access Service (SAS) of the Emergency Department of the CHG du Havre is a telephone regulation (i.e., orientation) service for users of Le Havre. Access to this service, during a call, gives access to a Medical Regulation Assistant (ARM) (first contact) who determines, in less than 30 seconds, the degree of urgency applicable to the "caller" in order to direct the latter to the "primary care" channel or the "urgent medical assistance" channel. Thus, in the context of a non-life-threatening emergency, this service allows access during the day to a consultation with a healthcare professional. When their primary care physician is not available, the "caller" is directed by a Medical Regulation Assistant (ARM) to an Unscheduled Care Operator (OSNP) who can provide medical advice, offer a teleconsultation, or direct them, depending on the situation, to an unscheduled care consultation in an office, at home, or at a health center. This service therefore allows for patient referrals and gives patients direct access to healthcare professionals known as "performers" of primary care (doctor, midwife, dentist) within very short timeframes (most often during the day, and 48 hours at the latest). This medical regulation is made possible through the use of a shared calendar between independent healthcare professionals and the healthcare access service (SAS). In the event of a life-threatening emergency, the "caller" is directed by the Medical Regulation Assistant (ARM) to an emergency Medical Regulation Assistant (ARM) who assesses the actual degree of urgency, the medical needs and the possibility of triggering the SAMU intervention. Before its implementation, the patient journey was complicated by the lack of a link between regulation and so-called "field" medical professionals, now called "performers" of primary care. Indeed, the initial so-called "standard" regulation system did not have a "primary care" referral system (with very rapid appointments to primary care for semi-emergencies (unscheduled community care)), potentially saving recourse to emergency services or medical time in situations not requiring medical advice (request for contact details of on-call pharmacy).

DETAILED DESCRIPTION:
The SAS represents an evolution of SAMU medical regulation, no longer based solely on emergency medical assistance (the standard regulation system), but also combining it with outpatient medical regulation.

It is therefore a multi-professional platform that saves medical time by delegating some of the tasks (pre-triage, administrative information gathering², scheduling unscheduled care appointments) to non-medical personnel specifically trained for the task (Unscheduled Care Operators (OSNP)). This study seeks to assess the benefits of this new system in a context of very high social expectations. A comparative assessment is necessary between the Emergency Department's Access to Care Service (SAS) and the former "standard" regulation system to understand the overall impact of the "SAS" on the Le Havre healthcare area.

This study has multiple perspectives:

* For users, the aim is to compare the care trajectory of regulated users (healthcare professional(s) seen, emergency room stay, hospitalization, etc.) by the "SAS" versus "standard" regulation and to understand the use of Unscheduled Care (SNP) provided in the Le Havre area;
* To assess the medical-economic impact of the "SAS" versus "standard" regulation.
* For healthcare professionals, it is a question of understanding and describing the interactions between the "effectors" of primary care (doctor, midwife, dentist) and the regulators involved (Unscheduled Care Operator (OSNP) (via the Medical Regulation Assistant (ARM))) in the "SAS"

ELIGIBILITY:
Inclusion Criteria:

* For the primary analysis and secondary outcome measure 1:

  * All calls to 116-117 or 15 in the Le Havre area over the 40 study periods,
  * Non-opposition. Patients with a life-threatening emergency will be included in the primary analysis, even though there will be no pseudo-randomization of the systems for them. They are therefore included in the study.
* For the secondary analysis on patient compliance with the referral given by the regulating physician (secondary objective 2):

  * Non-opposition of patients who used the SNP call for the primary analysis,
  * Randomly selected by sampling calls to 116-117 or 15 made over the study periods defined by the protocol.
* For the qualitative component:

  * Major,
  * No opposition from regulators and major effectors of the SAS
  * Or No opposition from adult health patients in the Le Havre area who have used the unscheduled care system (outpatient or inpatient).

Exclusion Criteria:

* For the primary analysis and secondary objective 1:

  * Refusal to participate,
  * Non-French speaking.
* For the secondary analysis on patient compliance with the referral given by the regulating physician (secondary objective 2) and for the qualitative component:

  * Minor caller
  * Refusal to participate (patient or caller or both),
  * Non-French speaking (caller)
  * Only for adult healthcare users in the Le Havre area included in the qualitative component: Not having the independent capacity to use the SNP. Non-use of the SAS will not be a criterion for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Users of the health system: The concept of users applies not only to the sick person and their loved ones but, more broadly, to any actual or potential user of the health system, in the health and medico-social fields, in establishments as well as in outpatient care or in home care
Sampling Method: Probability Sample
Enrollment: 9280 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the savings in emergency room use attributable to the regulation system integrating the SAS compared to the standard control device | day 7
  Assessment of referral to an emergency department by the regulating physician who treated the patient (with or without urgent medical transport) by telephone call.

SECONDARY OUTCOMES:
Description of the guidance given by the regulating physician in each of the devices (secondary judgment criterion no. 1) | Day 7
  The patient's orientation following the call (medical advice) will be recorded and evaluated.
Description of the guidance given by the regulating physician in each of the devices (secondary judgment criterion no. 1) | Day 7
  The patient's orientation following the call (appointment with a healthcare professional) will be recorded and evaluated.
Assessment of the patient's compliance rate with the guidance given by the regulating physician (secondary judgment criterion no. 2) | Day 7
  The patient's compliance with the guidance given by the private regulating physician will be recorded and evaluated.
Assessment of the patient's compliance rate with the guidance given by the regulating physician (secondary judgment criterion no. 2) | Day 7
  The patient's compliance with the guidance given by the hospital regulating physician will be recorded and evaluated.
Evaluation of the medical-economic impact of "SAS" regulation versus "standard" regulation (Qualitative component) | Year 5
  Analysis of the budgetary impact, i.e. the difference in costs between the two systems, taking into account the direction indicated and the general degree of compliance with the directions from the point of view of health insurance over 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Le Havre Hospital Group,, Le Havre, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.